CLINICAL TRIAL: NCT05887908
Title: A Phase 3, Multi-Center, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Cefepime/Nacubactam or Aztreonam/Nacubactam Compared to Imipenem/Cilastatin in the Treatment of Complicated Urinary Tract Infections or Acute Uncomplicated Pyelonephritis, in Adults
Brief Title: Efficacy and Safety of Cefepime/Nacubactam or Aztreonam/Nacubactam Compared to Imipenem/Cilastatin in Subjects With Complicated Urinary Tract Infections or Acute Uncomplicated Pyelonephritis
Acronym: Integral-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OP0595-5
Record Dates: First submitted 2023-04-25; First posted 2023-06-05 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis; cUTI; AP
Keywords: OP0595; nacubactam; Integral
MeSH Terms: interventions — nacubactam; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- co-administration of cefepime and nacubactam (Experimental): co-administration of 2 g cefepime and 1 g nacubactam q8h (60 min. infusion)
  Interventions: Drug: co-administration of cefepime and nacubactam
- co-administration of aztreonam and nacubactam (Experimental): co-administration of 2 g aztreonam and 1 g nacubactam q8h (60 min. infusion)
  Interventions: Drug: co-administration of aztreonam and nacubactam
- imipenem/cilastatin (Active Comparator): combination of 1 g imipenem/1 g cilastatin q8h (60 min. infusion)
  Interventions: Drug: imipenem/cilastatin

INTERVENTIONS:
Drug: co-administration of cefepime and nacubactam — 2 g cefepime and 1 g nacubactam
  Arms: co-administration of cefepime and nacubactam
Drug: co-administration of aztreonam and nacubactam — 2 g aztreonama and 1 g nacubactam
  Arms: co-administration of aztreonam and nacubactam
Drug: imipenem/cilastatin — 1 g imipenem/1 g cilastatin
  Arms: imipenem/cilastatin

SUMMARY:
Phase 3 study to evaluate the efficacy and safety of cefepime/nacubactam or aztreonam/nacubactam compared to imipenem/cilastatin in the treatment of complicated urinary tract infections (cUTI) or acute uncomplicated pyelonephritis (AP).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least18 years of age (or age of legal consent, whichever is older) at the time of obtaining informed consent and who can be hospitalized throughout the Treatment Period;
2. Weight at most 140 kg;
3. Expectation, in the opinion of the Investigator, that the patient's cUTI or AP will require treatment with at least 5 days of IV antibiotics;

Exclusion Criteria:

1. Has a known imipenem- and/or meropenem-resistant Gram-negative uropathogen (at least 10^5 CFU/mL), isolated from study-qualifying urine culture; Note: If after randomization the susceptibility testing indicates resistance to imipenem and/or meropenem, the patient may remain on the study drug at the Investigator's discretion.
2. Has known or suspected single or concurrent infection with Acinetobacter spp. or other organisms that are not adequately covered by the study drug (eg, concurrent viral, mycobacterial, or fungal infection) and needs to be managed with other anti-infectives; Note: Patients with qualifying pathogen coinfected with a Gram-positive pathogen may be administered narrow spectrum, open-label glycopeptide (eg, vancomycin), oxazolidinone (eg, linezolid), or daptomycin concomitantly with the study drug at the Investigator's discretion.
3. Has only a known Gram-positive primary uropathogen (at least 10^5 CFU/mL), isolated from study qualifying urine culture;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- Bulgaria (4):
  - Meiji Research Site, Pleven
  - Meiji Research Site, Rousse
  - Meiji Research Site, Silistra
  - Meiji Research Site, Sofia
- China (19):
  - Meiji Research Site, Beijing
  - Meiji Research Site, Changchun
  - Meiji Research Site, Chongqing
  - Meiji Research Site, Fuyang
  - Meiji Research Site, Ganzhou
  - Meiji Research Site, Huaian
  - Meiji Research Site, Huzhou
  - Meiji Research Site, Nanchang
  - Meiji Research Site, Nanning
  - Meiji Research Site, Quanzhou
  - Meiji Research Site, Shanghai
  - Meiji Research Site, Shantou
  - Meiji Research Site, Shijiazhuang
  - Meiji Research Site, Taian
  - Meiji Research Site, Tianjin
  - Meiji Research Site, Xuancheng
  - Meiji Research Site, Yunnan
  - Meiji Research Site, Zhejiang
  - Meiji Research Site, Zhengzhou
- Czechia (4):
  - Meiji Research Site, Hradec Králové
  - Meiji Research Site, Liberec
  - Meiji Research Site, Prague
  - Meiji Research Site, Ústí nad Labem
- Estonia (4):
  - Meiji Research Site, Meegomäe, Võrumaa
  - Meiji Research Site, Kohtla-Järve
  - Meiji Research Site, Tallinn
  - Meiji Research Site, Tartu
- Georgia (3):
  - Meiji Research Site, Kutaisi
  - Meiji Research Site, Rustavi
  - Meiji Research Site, Tbilisi
- Japan (20):
  - Meiji Research Site, Fukuyama
  - Meiji Research Site, Gifu
  - Meiji Research Site, Ibaraki-Town, Higashiibaraki-County
  - Meiji Research Site, Iwakuni
  - Meiji Research Site, Kanazawa
  - Meiji Research Site, Kawachi-Nagano
  - Meiji Research Site, Kofu
  - Meiji Research Site, Kumamoto
  - Meiji Research Site, Matsumoto
  - Meiji Research Site, Mizumaki-Town, Onga-County
  - Meiji Research Site, Nagasaki
  - Meiji Research Site, Nankoku
  - Meiji Research Site, Ōita
  - Meiji Research Site, Ōtake
  - Meiji Research Site, Sagamihara
  - Meiji Research Site, Sapporo
  - Meiji Research Site, Shinjuku-ku
  - Meiji Research Site, Toyota
  - Meiji Research Site, Ueda
  - Meiji Research Site, Yokohama
- Latvia (2):
  - Meiji Research Site, Riga
  - Meiji Research Site, Valmiera
- Lithuania (2):
  - Meiji Research Site, Kaunas
  - Meiji Research Site, Vilnius
- Slovakia (3):
  - Meiji Research Site, Galanta
  - Meiji Research Site, Rimavská Sobota
  - Meiji Research Site, Svidník

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 678 patients were screened at 66 sites in 9 countries and 614 patients were radomized.
Groups:
- Cefepime/Nacubactam: 2 g cefepime/1 g nacubactam every 8 hours for at least 5 days and up to 14 days via IV infusion over a period of 60 minutes
- Aztreonam/Nacubactam: 2 g aztreonam/1 g nacubactam every 8 hours for at least 5 days and up to 14 days via IV infusion over a period of 60 minutes
- Imipenem/Cilastatin: 1 g imipenem/1 g cilastatin every 8 hours for at least 5 days and up to 14 days via IV infusion over a period of 60 minutes
Period: Overall Study
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Started | 309 | 154 | 151
Treated | 307 | 152 | 151
Completed Study Drug | 290 | 147 | 143
Completed | 284 | 144 | 139
Not Completed | 25 | 10 | 12
Not completed — Adverse Event | 6 | 1 | 1
Not completed — Physician Decision | 4 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 3
Not completed — Ineligibility after the start of the study | 4 | 1 | 0
Not completed — Subject non-compliance | 4 | 0 | 4
Not completed — Grew only a Gram-negative organism resistant to imipenem and/or meropenem | 0 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Required Use of Prohibited Concomitant Medications | 1 | 0 | 0
Not completed — Significant prolongation of the QT/QTc interval | 0 | 1 | 0
Not completed — Other Reason | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Population: m-MITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin | Total
Number analyzed (Participants) | 214 | 112 | 105 | 431
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 99 | 42 | 41 | 182
  >=65 years | 115 | 70 | 64 | 249
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 51 | 49 | 203
  Male | 111 | 61 | 56 | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Customized: Asian-Japanese | 12 | 6 | 5 | 23
  Race, Customized: Asian-Chinese | 23 | 9 | 7 | 39
  Race, Customized: Asian-other | 0 | 1 | 0 | 1
  Race, Customized: White | 179 | 96 | 93 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (14.83) | 66.4 (14.04) | 65.5 (15.57) | 64.8 (14.83)
Age, Customized [Count of Participants; unit: Participants]
  Age, Customized: <65 years | 99 | 42 | 41 | 182
  Age, Customized: 65 - 74 Years | 62 | 36 | 32 | 130
  Age, Customized: >=75 years | 53 | 34 | 32 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity, Customized: Hispanic or Latino | 1 | 0 | 2 | 3
  Ethnicity, Customized: Not Hispanic or Latino | 212 | 112 | 103 | 427
  Ethnicity, Customized: Unknown | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 12 | 6 | 5 | 23
  China | 23 | 10 | 7 | 40
  Other | 179 | 96 | 93 | 368
Primary infection type collected in eCRF [Count of Participants; unit: Participants]
  Complicated Urinary Tract Infection (cUTI) | 137 | 76 | 73 | 286
  Acute Uncomplicated Pyelonephritis (AP) | 77 | 36 | 32 | 145
Creatinine Clearance (CrCl) at baseline [Mean (Standard Deviation); unit: mL/min] | 86.9 (34.94) | 87.8 (40.1) | 82.0 (32.43) | 85.9 (35.78)
Creatinine Clearance (CrCl) group [Count of Participants; unit: Participants]
  <30 | 1 | 3 | 0 | 4
  >=30 and <60 | 46 | 30 | 27 | 103
  >=60 and <90 | 77 | 30 | 44 | 151
  >=90 and <=240 | 88 | 49 | 33 | 170
  >240 | 0 | 0 | 0 | 0
  Data not collected for Creatinine Clearance (CrCl) at baseline | 2 | 0 | 1 | 3
Patients with secondary bacteremia at baseline [Count of Participants; unit: Participants]
  Yes | 15 | 9 | 10 | 34
  No | 199 | 103 | 95 | 397
Prior short-acting antibacterial therapy [Count of Participants; unit: Participants]
  Yes | 18 | 12 | 12 | 42
  No | 196 | 100 | 93 | 389

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieve Composite Clinical and Microbiological Success at TOC (Test of Cure Visit) in the Microbiological Modified Intent-to-Treat (m-MITT) Population
Description: Composite clinical and microbiological success is defined as the composite clinical outcome of cure and the microbiological outcome of eradication.
Time Frame: TOC (Test of Cure visit): 7 [±2] days after EOT (end of treatment) [Day 10 to 23 after the start of treatment]
Population: Microbiological Modified Intent-to-Treat (m-MITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 214 | 112 | 105
Participants | 176 | 81 | 64
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Test type: Non-Inferiority — Non-inferirority margin = 15.0%; If the lower limit of the 2-sided 95% CI of the group difference > -15.0%, non-inferiority is concluded. If non-inferiority is declared, a test for superiority will be performed. If the lower bound of the 95% CI > 0.0%, superiority will be declared; Difference in success proportion = 21.3, 95% CI 2-sided [10.9 to 32.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Test type: Non-Inferiority — Non-inferirority margin = 15.0%; If non-inferiority of the cefepime/nacubactam group is declared, a non-inferiority hypothesis test for the aztreonam/nacubactam group will be performed. For this analysis, the same approach as that used for the cefepime/nacubactam group will be used; Difference in success proportion = 11.4, 95% CI 2-sided [-1.2 to 23.7] — Miettinen-Nurminen confidence interval

2. Secondary Outcome: Proportion of Patients Who Achieve Composite Clinical and Microbiological Outcome
Description: Composite clinical and microbiological success is defined as the composite clinical outcome of cure and the microbiological outcome of eradication.
  Assessment of clinical outcome was based on Investigator's evaluation of the patient's clinical signs and symptoms, with cure defined as the complete resolution (or return to premorbid state) of the baseline signs and symptoms of cUTI or AP that were present at screening, such that no further antimicrobial therapy is warranted.
  Microbiological outcome was determined programmatically based on quantitative microbiological urine cultures, with eradication defined as the pathogen found at screening with 10^5 CFU/ml or more reduced to less than 10^3 CFU/ml.
  The results of subgroup analyses for only the two most frequent pathogens were shown because there were a large number of pathogen types, most of which were rare and sparsely represented in the dataset.
Time Frame: Outcome measurements were assessed at various visits: EA (Earlly Assessment): Day4, EOT (End of Treatment): Day5 to Day14, TOC (Test of Cure visit): Day10 to Day 23, FUP (Follow-Up visit): Day17 to Day30
Population: m-MITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 214 | 112 | 105
Participants
  Composite clinical and microbiological success at EA (Early Assessment visit) | 201 | 110 | 96
  Composite clinical and microbiological success at EOT (End of Treatment visit) | 199 | 102 | 94
  Composite clinical and microbiological success at FUP (Follow-up visit) | 147 | 73 | 65
  Composite clinical and microbiological success at TOC by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Composite clinical and microbiological success at TOC by baseline pathogen: Escherichia coli | 135 | 62 | 45
  Composite clinical and microbiological success at TOC by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Composite clinical and microbiological success at TOC by baseline pathogen: Klebsiella pneumoniae | 27 | 11 | 9
  Composite clinical and microbiological success at EOT by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Composite clinical and microbiological success at EOT by baseline pathogen: Escherichia coli | 151 | 81 | 66
  Composite clinical and microbiological success at EOT by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Composite clinical and microbiological success at EOT by baseline pathogen: Klebsiella pneumoniae | 30 | 10 | 16
  Composite clinical and microbiological success at FUP by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Composite clinical and microbiological success at FUP by baseline pathogen: Escherichia coli | 112 | 57 | 44
  Composite clinical and microbiological success at FUP by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Composite clinical and microbiological success at FUP by baseline pathogen: Klebsiella pneumoniae | 20 | 9 | 11
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EA; Test type: Other — Descriptive analysis; Difference in success proportion = 2.5, 95% CI 2-sided [-3.2 to 9.9] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EA; Test type: Other — Descriptive analysis; Difference in success proportion = 6.8, 95% CI 2-sided [1.1 to 14.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 3: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EOT; Test type: Other — Descriptive analysis; Difference in success proportion = 3.5, 95% CI 2-sided [-2.7 to 11.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 4: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EOT; Test type: Other — Descriptive analysis; Difference in success proportion = 1.5, 95% CI 2-sided [-6.6 to 10.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 5: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at FUP; Test type: Other — Descriptive analysis; Difference in success proportion = 6.8, 95% CI 2-sided [-4.1 to 18.1] — Miettinen-Nurminen confidence interval
Statistical Analysis 6: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at FUP; Test type: Other — Descriptive analysis; Difference in success proportion = 3.3, 95% CI 2-sided [-9.5 to 16.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 7: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at TOC by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 24.1, 95% CI 2-sided [12.0 to 36.6] — Miettinen-Nurminen confidence interval
Statistical Analysis 8: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at TOC by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 10.5, 95% CI 2-sided [-4.2 to 24.9] — Miettinen-Nurminen confidence interval
Statistical Analysis 9: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at TOC by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 28.1, 95% CI 2-sided [1.8 to 54.1] — Miettinen-Nurminen confidence interval
Statistical Analysis 10: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at TOC by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 35.4, 95% CI 2-sided [1.1 to 61.6] — Miettinen-Nurminen confidence interval
Statistical Analysis 11: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EOT by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 6.4, 95% CI 2-sided [-1.3 to 16.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 12: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EOT by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 4.2, 95% CI 2-sided [-5.6 to 14.7] — Miettinen-Nurminen confidence interval
Statistical Analysis 13: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EOT by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -6.3, 95% CI 2-sided [-20.3 to 13.9] — Miettinen-Nurminen confidence interval
Statistical Analysis 14: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at EOT by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -16.7, 95% CI 2-sided [-45.4 to 5.2] — Miettinen-Nurminen confidence interval
Statistical Analysis 15: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at FUP by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 11.2, 95% CI 2-sided [-1.7 to 24.4] — Miettinen-Nurminen confidence interval
Statistical Analysis 16: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at FUP by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 6.2, 95% CI 2-sided [-8.7 to 20.9] — Miettinen-Nurminen confidence interval
Statistical Analysis 17: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at FUP by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -6.3, 95% CI 2-sided [-31.9 to 23.1] — Miettinen-Nurminen confidence interval
Statistical Analysis 18: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Composite clinical and microbiological success at FUP by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 6.3, 95% CI 2-sided [-28.8 to 37.9] — Miettinen-Nurminen confidence interval

3. Secondary Outcome: Proportion of Patients With a Clinical Outcome of Cure
Description: Assessment of clinical outcome was based on Investigator's evaluation of the patient's clinical signs and symptoms, with cure defined as the complete resolution (or return to premorbid state) of the baseline signs and symptoms of cUTI or AP that were present at screening, such that no further antimicrobial therapy is warranted.
  The results of subgroup analyses for only the two most frequent pathogens were shown because there were a large number of pathogen types, most of which were rare and sparsely represented in the dataset.
Time Frame: as for outcome 2
Population: m-MITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 214 | 112 | 105
Participants
  Clinical outcome of cure at EA | 9 | 4 | 2
  Clinical outcome of cure at EOT | 204 | 106 | 100
  Clinical outcome of cure at TOC | 195 | 103 | 92
  Clinical outcome of cure at FUP | 188 | 98 | 89
  Clinical outcome of cure at EA by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Clinical outcome of cure at EA by baseline pathogen: Escherichia coli | 5 | 3 | 1
  Clinical outcome of cure at EA by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Clinical outcome of cure at EA by baseline pathogen: Klebsiella pneumoniae | 2 | 1 | 0
  Clinical outcome of cure at EOT by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Clinical outcome of cure at EOT by baseline pathogen: Escherichia coli | 155 | 84 | 71
  Clinical outcome of cure at EOT by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Clinical outcome of cure at EOT by baseline pathogen: Klebsiella pneumoniae | 31 | 11 | 16
  Clinical outcome of cure at TOC by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Clinical outcome of cure at TOC by baseline pathogen: Escherichia coli | 148 | 82 | 67
  Clinical outcome of cure at TOC by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Clinical outcome of cure at TOC by baseline pathogen: Klebsiella pneumoniae | 30 | 11 | 13
  Clinical outcome of cure at FUP by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Clinical outcome of cure at FUP by baseline pathogen: Escherichia coli | 143 | 78 | 62
  Clinical outcome of cure at FUP by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Clinical outcome of cure at FUP by baseline pathogen: Klebsiella pneumoniae | 28 | 11 | 15
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EA; Test type: Other — Descriptive analysis; Difference in success proportion = 2.3, 95% CI 2-sided [-2.8 to 6.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EA; Test type: Other — Descriptive analysis; Difference in success proportion = 1.7, 95% CI 2-sided [-3.5 to 7.2] — Miettinen-Nurminen confidence interval
Statistical Analysis 3: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EOT; Test type: Other — Descriptive analysis; Difference in success proportion = 0.1, 95% CI 2-sided [-4.6 to 6.4] — Miettinen-Nurminen confidence interval
Statistical Analysis 4: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EOT; Test type: Other — Descriptive analysis; Difference in success proportion = -0.6, 95% CI 2-sided [-7.1 to 6.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 5: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at TOC; Test type: Other — Descriptive analysis; Difference in success proportion = 3.5, 95% CI 2-sided [-3.3 to 11.8] — Miettinen-Nurminen confidence interval
Statistical Analysis 6: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at TOC; Test type: Other — Descriptive analysis; Difference in success proportion = 4.3, 95% CI 2-sided [-3.9 to 13.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 7: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at FUP; Test type: Other — Descriptive analysis; Difference in success proportion = 3.1, 95% CI 2-sided [-4.5 to 12.1] — Miettinen-Nurminen confidence interval
Statistical Analysis 8: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at FUP; Test type: Other — Descriptive analysis; Difference in success proportion = 2.7, 95% CI 2-sided [-6.6 to 12.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 9: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EA by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 1.8, 95% CI 2-sided [-4.2 to 6.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 10: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EA by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 2.1, 95% CI 2-sided [-4.1 to 8.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 11: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EA by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 6.3, 95% CI 2-sided [-13.9 to 20.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 12: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EA by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 8.3, 95% CI 2-sided [-12.6 to 36.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 13: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EOT by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 2.3, 95% CI 2-sided [-3.5 to 10.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 14: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EOT by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 1.0, 95% CI 2-sided [-6.9 to 9.6] — Miettinen-Nurminen confidence interval
Statistical Analysis 15: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EOT by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -3.1, 95% CI 2-sided [-15.9 to 16.8] — Miettinen-Nurminen confidence interval
Statistical Analysis 16: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at EOT by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -8.3, 95% CI 2-sided [-36.0 to 12.6] — Miettinen-Nurminen confidence interval
Statistical Analysis 17: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at TOC by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 3.2, 95% CI 2-sided [-4.5 to 13.1] — Miettinen-Nurminen confidence interval
Statistical Analysis 18: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at TOC by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 4.0, 95% CI 2-sided [-5.3 to 14.2] — Miettinen-Nurminen confidence interval
Statistical Analysis 19: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at TOC by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 12.5, 95% CI 2-sided [-6.0 to 38.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 20: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at TOC by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 10.4, 95% CI 2-sided [-20.5 to 37.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 21: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at FUP by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 6.7, 95% CI 2-sided [-2.6 to 17.8] — Miettinen-Nurminen confidence interval
Statistical Analysis 22: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at FUP by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 6.1, 95% CI 2-sided [-5.0 to 17.8] — Miettinen-Nurminen confidence interval
Statistical Analysis 23: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at FUP by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -6.3, 95% CI 2-sided [-23.6 to 17.6] — Miettinen-Nurminen confidence interval
Statistical Analysis 24: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Clinical outcome of cure at FUP by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -2.1, 95% CI 2-sided [-30.9 to 22.3] — Miettinen-Nurminen confidence interval

4. Secondary Outcome: Proportion of Patients With a Microbiological Outcome of Eradication
Description: Microbiological outcome was determined programmatically based on quantitative microbiological urine cultures, with eradication defined as the pathogen found at screening with 10^5 CFU/ml or more reduced to less than 10^3 CFU/ml.
  The results of subgroup analyses for only the two most frequent pathogens were shown because there were a large number of pathogen types, most of which were rare and sparsely represented in the dataset.
Time Frame: as for outcome 2
Population: m-MITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 214 | 112 | 105
Participants
  Microbiological outcome of eradication at EA | 205 | 112 | 97
  Microbiological outcome of eradication at EOT | 203 | 105 | 95
  Microbiological outcome of eradication at TOC | 184 | 83 | 67
  Microbiological outcome of eradication at FUP | 157 | 75 | 68
  Microbiological outcome of eradication at EA by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Microbiological outcome of eradication at EA by baseline pathogen: Escherichia coli | 155 | 89 | 71
  Microbiological outcome of eradication at EA by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Microbiological outcome of eradication at EA by baseline pathogen: Klebsiella pneumoniae | 30 | 12 | 13
  Microbiological outcome of eradication at EOT by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Microbiological outcome of eradication at EOT by baseline pathogen: Escherichia coli | 154 | 83 | 67
  Microbiological outcome of eradication at EOT by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Microbiological outcome of eradication at EOT by baseline pathogen: Klebsiella pneumoniae | 30 | 11 | 16
  Microbiological outcome of eradication at TOC by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Microbiological outcome of eradication at TOC by baseline pathogen: Escherichia coli | 141 | 63 | 47
  Microbiological outcome of eradication at TOC by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Microbiological outcome of eradication at TOC by baseline pathogen: Klebsiella pneumoniae | 27 | 11 | 10
  Microbiological outcome of eradication at FUP by baseline pathogen: Escherichia coli: number analyzed (Participants) | 162 | 89 | 76
  Microbiological outcome of eradication at FUP by baseline pathogen: Escherichia coli | 119 | 58 | 46
  Microbiological outcome of eradication at FUP by baseline pathogen: Klebsiella pneumoniae: number analyzed (Participants) | 32 | 12 | 16
  Microbiological outcome of eradication at FUP by baseline pathogen: Klebsiella pneumoniae | 22 | 9 | 12
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EA; Test type: Other — Descriptive analysis; Difference in success proportion = 3.4, 95% CI 2-sided [-1.7 to 10.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EA; Test type: Other — Descriptive analysis; Difference in success proportion = 7.6, 95% CI 2-sided [3.9 to 14.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 3: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EOT; Test type: Other — Descriptive analysis; Difference in success proportion = 4.4, 95% CI 2-sided [-1.3 to 11.9] — Miettinen-Nurminen confidence interval
Statistical Analysis 4: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EOT; Test type: Other — Descriptive analysis; Difference in success proportion = 3.3, 95% CI 2-sided [-4.2 to 11.2] — Miettinen-Nurminen confidence interval
Statistical Analysis 5: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at TOC; Test type: Other — Descriptive analysis; Difference in success proportion = 22.2, 95% CI 2-sided [12.2 to 32.7] — Miettinen-Nurminen confidence interval
Statistical Analysis 6: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at TOC; Test type: Other — Descriptive analysis; Difference in success proportion = 10.3, 95% CI 2-sided [-2.0 to 22.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 7: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at FUP; Test type: Other — Descriptive analysis; Difference in success proportion = 8.6, 95% CI 2-sided [-2.0 to 19.7] — Miettinen-Nurminen confidence interval
Statistical Analysis 8: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at FUP; Test type: Other — Descriptive analysis; Difference in success proportion = 2.2, 95% CI 2-sided [-10.4 to 14.8] — Miettinen-Nurminen confidence interval
Statistical Analysis 9: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EA by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 2.3, 95% CI 2-sided [-3.5 to 10.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 10: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EA by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 6.6, 95% CI 2-sided [2.3 to 14.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 11: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EA by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 12.5, 95% CI 2-sided [-6.0 to 38.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 12: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EA by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 18.8, 95% CI 2-sided [-8.3 to 43.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 13: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EOT by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 6.9, 95% CI 2-sided [-0.1 to 16.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 14: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EOT by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 5.1, 95% CI 2-sided [-3.9 to 15.1] — Miettinen-Nurminen confidence interval
Statistical Analysis 15: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EOT by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -6.3, 95% CI 2-sided [-20.3 to 13.9] — Miettinen-Nurminen confidence interval
Statistical Analysis 16: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at EOT by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -8.3, 95% CI 2-sided [-36.0 to 12.6] — Miettinen-Nurminen confidence interval
Statistical Analysis 17: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at TOC by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 25.2, 95% CI 2-sided [13.5 to 37.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 18: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at TOC by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 8.9, 95% CI 2-sided [-5.5 to 23.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 19: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at TOC by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 21.9, 95% CI 2-sided [-3.4 to 48.5] — Miettinen-Nurminen confidence interval
Statistical Analysis 20: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at TOC by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 29.2, 95% CI 2-sided [-4.4 to 56.0] — Miettinen-Nurminen confidence interval
Statistical Analysis 21: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at FUP by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 12.9, 95% CI 2-sided [0.3 to 25.9] — Miettinen-Nurminen confidence interval
Statistical Analysis 22: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at FUP by baseline pathogen: Escherichia coli; Test type: Other — Descriptive analysis; Difference in success proportion = 4.6, 95% CI 2-sided [-10.1 to 19.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 23: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at FUP by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = -6.3, 95% CI 2-sided [-30.4 to 22.6] — Miettinen-Nurminen confidence interval
Statistical Analysis 24: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Microbiological outcome of eradication at FUP by baseline pathogen: Klebsiella pneumoniae; Test type: Other — Descriptive analysis; Difference in success proportion = 0.0, 95% CI 2-sided [-34.0 to 31.5] — Miettinen-Nurminen confidence interval

5. Secondary Outcome: Proportion of Patients With a Clinical Outcome of Cure at TOC in Patients With Secondary Bacteremia at Baseline
Description: Patients with isolation of a gram-negative bacteria from at least 1 blood culture at baseline and this isolated pathogen is also identified from the site of infection and signs and symptoms of secondary bacteremia were determined programmatically as secondary bacteremia.
  Assessment of clinical outcome was based on signs and symptoms, with cure defined as complete resolution or significant improvement of the baseline signs and symptoms of secondary bacteremia.
Time Frame: TOC (Test of Cure visit): Day 10 to Day 23 after the start of treatment
Population: Patients with secondary bacteremia at baseline in m-MITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 15 | 9 | 10
Participants | 12 | 8 | 6
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Descriptive analysis; Difference in success proportion = 20.0, 95% CI 2-sided [-16.0 to 54.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Descriptive analysis; Difference in success proportion = 28.9, 95% CI [-13.0 to 62.1] — Miettinen-Nurminen confidence interval

6. Secondary Outcome: Proportion of Patients With a Microbiological Outcome of Eradication at TOC in Patients With Secondary Bacteremia at Baseline
Description: Patients with isolation of a gram-negative bacteria from at least 1 blood culture at baseline and this isolated pathogen is also identified from the site of infection and signs and symptoms of secondary bacteremia were determined programmatically as secondary bacteremia.
  Microbiological outcome will be determined programmatically based on blood cultures, with eradication defined as the pathogen found at screening is negative in blood culture.
Time Frame: TOC (Test of Cure visit): Day 10 to Day 23 after the start of treatment
Population: Patients with secondary bacteremia at baseline in m-MITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 15 | 9 | 10
Participants | 12 | 8 | 6
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Descriptive analysis; Difference in success proportion = 20.0, 95% CI 2-sided [-16.0 to 54.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Descriptive analysis; Difference in success proportion = 28.9, 95% CI [-13.0 to 62.1] — Miettinen-Nurminen confidence interval

7. Secondary Outcome: Proportion of Patients Who Are Free From the Definition of Secondary Bacteremia AND a Clinical Outcome of Cure AND a Microbiological Outcome of Eradication From cUTI or AP at TOC in Patients With Secondary Bacteremia at Baseline
Description: Patients with isolation of a gram-negative bacteria from at least 1 blood culture at baseline and this isolated pathogen is also identified from the site of infection and signs and symptoms of secondary bacteremia were determined programmatically as secondary bacteremia. For cUTI/AP,Assessment is done by the same way as "Proportion of patients who achieve composite clinical and microbiological outcome". For secondary bacteremia, assessment of clinical outcome was based on signs and symptoms, with cure defined as complete resolution or significant improvement of the baseline signs and symptoms of secondary bacteremia. Microbiological outcome will be determined programmatically based on blood cultures, with eradication defined as the pathogen found at screening is negative in blood culture.
Time Frame: TOC (Test of Cure visit): Day 10 to Day 23 after the start of treatment
Population: Patients with secondary bacteremia at baseline in m-MITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 15 | 9 | 10
Participants | 11 | 4 | 2
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Desriptive analysis; Difference in success proportion = 53.3, 95% CI 2-sided [12.8 to 78.1] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Descriptive analysis; Difference in success proportion = 24.4, 95% CI 2-sided [-18.4 to 60.5] — Miettinen-Nurminen confidence interval

8. Secondary Outcome: Proportion of Patients Who Are Free From Secondary Bacteremia in Patients With Secondary Bacteremia at TOC
Description: Patients with isolation of a gram-negative bacteria from at least 1 blood culture at baseline and this isolated pathogen is also identified from the site of infection and signs and symptoms of secondary bacteremia were determined programmatically as secondary bacteremia. Assessment of clinical outcome was based on signs and symptoms, with cure defined as complete resolution or significant improvement of the baseline signs and symptoms of secondary bacteremia. Microbiological outcome will be determined programmatically based on blood cultures, with eradication defined as the pathogen found at screening is negative in blood culture.
Time Frame: TOC (Test of Cure visit): Day 10 to Day 23 after the start of treatment
Population: Patients with secondary bacteremia at baseline in m-MITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
Number analyzed (Participants) | 15 | 9 | 10
Participants | 12 | 8 | 6
Statistical Analysis 1: Comparison: Cefepime/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Descriptive analysis; Difference in success proportion = 20.0, 95% CI 2-sided [-16.0 to 54.3] — Miettinen-Nurminen confidence interval
Statistical Analysis 2: Comparison: Aztreonam/Nacubactam vs Imipenem/Cilastatin; Test type: Other — Descriptive analysis; Difference in success proportion = 28.9, 95% CI 2-sided [-13.0 to 62.1] — Miettinen-Nurminen confidence interval

ADVERSE EVENTS:
Time Frame: Up to follow-up visit (maximum Day 30)
Arm/Group | Cefepime/Nacubactam | Aztreonam/Nacubactam | Imipenem/Cilastatin
All-Cause Mortality (participants affected / at risk) | 1/306 | 0/152 | 0/150
Serious Adverse Events (participants affected / at risk) | 6/306 | 4/152 | 5/150
Other Adverse Events (participants affected / at risk) | 100/306 | 45/152 | 65/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cefepime/Nacubactam (N=306) | Aztreonam/Nacubactam (N=152) | Imipenem/Cilastatin (N=150)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cefepime/Nacubactam (N=306) | Aztreonam/Nacubactam (N=152) | Imipenem/Cilastatin (N=150)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 3 (3) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 10 (10)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Asymptomatic bacteriuria (Infections and infestations) | 3 (3) | 7 (7) | 5 (5)
Headache (Nervous system disorders) | 10 (11) | 8 (8) | 6 (6)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 5 (5) | 3 (3) | 0 (0)
Any AEs with frequency less than 2% (General disorders) | 42 (42) | 13 (13) | 17 (17)

LIMITATIONS AND CAVEATS:
The analysis plan included subgroup analyses by pathogen for some secondary endpoints. However, there were a large number of pathogen types, most of which were rare and sparsely represented in the dataset. Therefore, we present the results of subgroup analyses for only the two most frequent pathogens, as analyses for the others were considered statistically unreliable and clinically uninformative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The following contract has been concluded with the sites in the clinical trial agreement:

* Information obtained from the results of the trial must not be leaked without the Sponsor's prior written consent.
* If information obtained from the trial is to be published outside the institution, such as at an academic conference, prior written consent must be obtained from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT05887908/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT05887908/SAP_001.pdf